CLINICAL TRIAL: NCT02377804
Title: Changes in Spasticity, Range of Motion and Pressure Pain Sensitivity in Patients With Stroke After the Application of Dry Needling in the Shoulder Musculature
Brief Title: Dry Needling for Spasticity in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HBMA-URJC
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: dry needling; spasticity; pain
MeSH Terms: conditions — Stroke; Muscle Spasticity; Pain | interventions — Dry Needling; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental intervention (Experimental): The experimental intervention will consist of 3 sessions, one per week, of 45min of physical therapy including mobilizations of the scapular region, manual therapies targeted to decrease muscle tone, neuromodulatory techniques for spasticity and proprioceptive exercises for the upper extremity. In addition, during this intervention patients will also receive deep dry needling with disposable stainless steel needles (0.3mm x 50mm) that will be inserted into the skin over taut bands of the spastic musculature of the shoulder area: upper trapezius, subscapularis, infraspinatus, and pectoralis mayor
  Interventions: Other: Dry needling; Other: Physical Therapy; Device: stainless steel needles (0.3mm x 50mm)
- Control intervention (Active Comparator): The control intervention will consist of 3 sessions, one per week, of 45min of physical therapy including mobilizations of the scapular region, manual therapies targeted to decrease muscle tone, neuromodulatory techniques for spasticity and proprioceptive exercises for the upper extremity.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Dry needling — Patients will receive deep dry needling with disposable stainless steel needles (0.3mm x 50mm) that will be inserted into the skin over taut bands of the spastic musculature of the shoulder area: upper trapezius, subscapularis, infraspinatus, and pect
  Arms: Experimental intervention
Other: Physical Therapy — Patients will receive 3 sessions, one per week, of 45min of physical therapy including mobilizations of the scapular region, manual therapies targeted to decrease muscle tone, neuromodulatory techniques for spasticity and proprioceptive exercises for the upper extremity
Device: stainless steel needles (0.3mm x 50mm)
  Arms: Experimental intervention

SUMMARY:
Stroke is the leading cause of physical disability due to the presence of spasticity. Different needling techniques, including Botulinum Toxin A are proposed for management of spasticity; however results are conflicting. The presence of spasticity in the upper extremity implies several impairments for daily life activities. No study has investigated the effects of deep dry needling inserted into the targeted spastic musculature of the shoulder region in patients who had suffered a stroke. The investigators will conduct a randomized controlled trial investigating the effects of the inclusion of deep dry needling into a rehabilitation program over the musculature of the shoulder region, pressure pain hyperalgesia and range of motion in individuals with chronic stroke. The investigators hypothesize that patients receiving dry needling into the spastic shoulder musculature would exhibit greater improvements in spasticity, pressure sensitivity and range of motion than those who will not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* first-ever unilateral stroke;
* hemiplegia resulting from stroke;
* age between 40 and 65 years old;
* presence of hypertonicity in the upper extremity;
* restricted range of motion of the shoulder

Exclusion Criteria:

* recurrent stroke;
* previous treatment with nerve blocks, motor point injections with neurolytic agents for spasticity at any time;
* previous treatment with BTX-A in the 6 months prior the study;
* severe cognitive deficits; 5, progressive or severe neurologic diseases, e.g., heart conditions, unstable hypertension, fracture or implants in the lower extremity;
* fear to needles;
* any contraindication for deep dry needling, e.g., anticoagulants, infections, bleeding, or psychotic.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in spasticity before and after the intervention | Baseline and immediate after the interventionBaseline (1 week before) and 1 week after intervention
  Spasticity in the affected ankle joint will be evaluated with the Modified Modified Ashworth Scale (MMAS). The examiner passively moved the upper extremity in a stretching direction of each muscle (shoulder depression, shoulder external rotation, shoulder internal rotation, and shoulder abduction 90º combined with external rotation, respectively), back and forth at least 5 times and evaluated the degree of resistance to the movement on a scale from 0-4

SECONDARY OUTCOMES:
Changes in pressure pain sensitivity before and after the intervention | Baseline (1 week before) and 1 week after intervention
  Pressure pain thresholds, defined as the amount of pressure applied for the pressure sensation to first change to pain, will be assessed with a mechanical pressure algometer (Pain Diagnosis and Treatment Inc, New York, USA) unilaterally over the affected infraspinatus and deltoid muscles and bilaterally over the C5/C6 zygapophyseal joint.
Changes in shoulder mobility before and after the intervention | Baseline (1 week before) and 1 week after intervention
  A universal goniometer will be used to determine the participant's shoulder range of motion in flexion, abduction and external rotation

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, Study Director — Universidad Rey Juan Carlos
Locations (2):
- Spain (2):
  - Universidad Rey Juan Carlos, Alcorcón, Madrid
  - Hospital Beta María Ana, Madrid, Madrid